CLINICAL TRIAL: NCT04476667
Title: Online Delivery of Psychotherapy, Tailored to Patients' Suffering from Mental Health Problems Due to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-683-20
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Issue; Covid19; Anxiety Disorders; Depression
Keywords: Anxiety; Depression; COVID-19; Online Psychotherapy; Mental Health
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants selected for the e-psychotherapy group will receive a 9-week program that includes a combination of CBT, mindfulness, and problem-based therapy, in addition to TAU. The control group will receive treatment as usual during the first 9 weeks; if they still present significant symptoms (less than 50% response to treatment from baseline), they will be offered the e-psychotherapy program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- e-Psychotherapy (Experimental): Participants will receive a 9-week program with CBT, mindfulness, and problem-based therapy, in addition to TAU. The content will be customized to reflect challenges faced through the COVID-19 pandemic and developed into interactive and engaging modules. All sessions and interactions will occur through Online Psychotherapy Tool (OPTT), a secure online platform. Participants will be assigned to a team of psychiatrists and social workers (SWs). The SW working with each patient will assign a pre-designed therapy module to that patient on a specific day of the week through OPTT. Participants will then be able to access the therapy content at any time throughout the week. Each module will highlight a different topic and include general information, an overview of skills, and homework that is to be completed by a specific day that week. This homework will be directly submitted through OPTT to the clinician who will provide personalized feedback to the patient.
  Interventions: Behavioral: e-Psychotherapy
- Treatment as Usual (No Intervention): The control group will receive treatment as usual during the first 9 weeks; if they still present significant symptoms (less than 50% response to treatment from baseline), they will be offered the e-psychotherapy program.

INTERVENTIONS:
Behavioral: e-Psychotherapy — Module Content: The first 3 sessions will be designed to address the symptoms caused by fear of illness or concerns about personal safety in the context of pandemic. Electronic-CBT (e-CBT) modules will focus on problem solving techniques, with mindfulness practices included, to help build healthy coping skills to address the uncertainties surrounding the COVID-19 pandemic. e-CBT modules will involve guiding participants to develop constructive and balanced coping strategies through 5 focuses: stimulus control, cognitive therapy, sleep hygiene, relaxation therapy, and sleep restriction. Additional focus will be placed on the connection between thoughts, behaviours, emotions, physical reaction and one's environment.
  Arms: e-Psychotherapy

SUMMARY:
The recent COVID-19 pandemic has affected many aspects of individuals social life and its negative consequences on Canadian public health go far beyond the direct overload of the hospital care system. Self-isolation and financial uncertainty can significantly deteriorate individuals' mental health, which is only going to aggravate with prolonged physical distancing strategies. Adding to this is the personal and public trauma of lost lives and soon there will be an unprecedented epidemic of mental health problems with crushing effects on the public health sector and economy. To meet this huge new demand for an already strained health system, there is a need for innovative new approaches that significantly expand the capacity of care delivery. While it may not be possible in the short term to increase the number of mental healthcare providers or the number of hours they work, improving their time spent efficiently might be the solution. Virtual care and online delivery of psychotherapy, shown to be clinically effective, efficient and cost-effective, might be the perfect solution to address the high demand faced now. The investigators aim to establish the first academic online psychotherapy clinic to manage mental health problems secondary to COVID-19. The goal is to evaluate the feasibility and efficacy of treating COVID-19 related mental health issues in this clinic, offering a 10-week, diagnosis-specific, online psychotherapy program. The investigators will use the Online Psychotherapy Tool (OPTT), a secure cloud-based digital mental health platform, developed by the PI, Dr. Alavi. Potentially, this method of care delivery could increase care capacity by four-folds. The findings from this project have the potential to influence clinical practice and policy and increase accessibility to care during COVID-19 pandemic, without sacrificing the quality of care.

DETAILED DESCRIPTION:
Participants: Participants (n=80) aged 18-65 years will be recruited from referrals within the outpatient clinics of HDH and PCH. Participants who consent to take part in the study will be evaluated by one of the psychiatrists on the team through a video appointment. Diagnosis of MDD and/or GAD will be confirmed using the DSM-5 and approved through the M.I.N.I. The inclusion criteria for the study will include the capacity to consent; a diagnosis of MDD and/or GAD, the ability to speak and read English, and having consistent and reliable access to the internet. Exclusion criteria include active psychosis, acute mania, severe alcohol or substance use disorder, and/or active suicidal or homicidal ideation. If a participant is receiving another form of psychotherapy, they will also be excluded from the study. If eligible for the study, participants will be randomly assigned to either the electronic psychotherapy (e-psychotherapy) or control (i.e. Treatment as usual (TAU)) group, stratified by sex, age group, and gender.

Participants selected for the e-psychotherapy group will receive a 9-week program that includes a combination of CBT, mindfulness, and problem-based therapy, in addition to TAU. The content of the e-psychotherapy program will be customized to reflect the challenges that individuals face through the COVID-19 pandemic and will be developed into interactive and engaging therapy modules. All online sessions and interactions will occur through Online Psychotherapy Tool (OPTT), a secure online platform.

Through OPTT, all participants will be assigned to a team of psychiatrists and social workers (SWs). The SW working with each patient will assign a pre-designed therapy module to that patient on a specific day of the week through OPTT. Participants will then be able to access the therapy content at any time throughout the week. Each weekly module will highlight a different topic and include general information, an overview of skills, and homework that is to be completed by a specific day that week. Completing each weekly module requires an average time commitment of 40-minutes, which can be completed at once or in blocks of time. This homework will be directly submitted through OPTT to the clinician who will then provide personalized feedback to the patient. To ensure a consistent high-quality outcome, SWs will use pre-designed session-specific feedback templates to respond to each weekly patient submission. Each patient's care team will be able to securely communicate through OPTT to make decisions regarding each patient's care path. The control group will receive treatment as usual during the first 9 weeks; if they still present significant symptoms (less than 50% response to treatment from baseline), they will be offered the e-psychotherapy program.

Module Content: The first 3 sessions will be designed to address the symptoms caused by fear of illness or concerns about personal safety in the context of a pandemic. Electronic-CBT (e-CBT) modules will focus on problem-solving techniques, with mindfulness practices included, to help build healthy coping skills to address the uncertainties surrounding the COVID-19 pandemic. e-CBT modules will involve guiding participants to develop constructive and balanced coping strategies through 5 focuses: stimulus control, cognitive therapy, sleep hygiene, relaxation therapy, and sleep restriction. Additional focus will be placed on the connection between thoughts, behaviours, emotions, physical reaction and one's environment.

Training: Through training, all SWs will learn the standard care pathway, the aim, and the content of each therapeutic session. Moreover, they will be provided sample homework from a patient and asked to provide feedback. Feedback templates will vary from session to session and SWs will personalize each template for each patients' homework. Training will occur through webinars and exercises with feedback.

Outcome Evaluation: Primary outcomes measured will be stress level changes based on the DASS-21, resilience based on RS-14, and quality of life-based on Q-LES-Q. Additional measurements will be made based on participant diagnosis (PHQ9, MADRS, GAD7). All questionnaires will be collected directly through OPTT at baseline, session 6, after the final session, and at a 6-month follow up. Healthcare providers will be asked about the feasibility of providing the e-psychotherapy, how it compared to in-person psychotherapy with respect to time commitment, feelings of 'connectedness' to the participant, and any perceived benefits/drawbacks to e-psychotherapy. From focus groups, factors related to personal, social, and cultural factors (gender, sexuality, background, supportive resources, structural/social barriers, etc.) will be extracted using an Interpretive Phenomenological Analysis (IPA) approach.

Ethics and Data Privacy: All procedures have been submitted for approval of ethical compliance to the Queen's University Health Sciences and Affiliated Teaching Hospitals Research Ethics Board. Only the care providers involved in the care of the participant will have access to their chart. Patients will only be identifiable by an ID number on the OPTT platform and their real identity and consent forms will be stored locally in a locked file cabinet and destroyed 5 years after the study completion date. Only anonymized data will be provided to the analysis team members.

OPTT is HIPAA, PIPEDA and SOC-2 compliant and all servers and databases are hosted in AWS Canada cloud infrastructure which is managed by Medstack to assure all provincial and federal privacy and security regulations are met. OPTT will not collect any identifiable personal information or IP addresses for privacy purposes. OPTT will only collect anonymized metadata to improve its service quality and provide advanced analytics to the clinician team. All data is encrypted by OPTT and no employee has direct access to patient data. All encrypted backups are kept in the S3 storage that is dedicated to Queen's University.

Data Analysis: Repeated MANOVA will be used to evaluate treatment efficacy in changes in scores on the DASS-21, RS-14 & Q-LES-Q between the participant groups (TAU, anxiety, and depression), and changes within each specific diagnosis at four different time points. Thematic analysis will be applied to analyze survey questions in order to better capture experiences, acceptability and patient-centeredness of e-psychotherapy. Descriptive analysis of time spent by each care team member for individual participants to evaluate the cost efficiency of care delivery will occur.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent
* Diagnosis of MDD and/or GAD
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Active psychosis
* Acute mania
* Severe alcohol or substance use disorder
* Active suicidal or homicidal ideation
* Participant receiving another form of psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Stress | Baseline, week 6, week 12
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) - Scale: 0-3 (0 = never, 3 = frequently)
Change in Resilience | Baseline, week 6, week 12
  14 Item Resilience Scale (RS-14) - Scale: 1-7 (1 = strongly disagree, 7 = strongly agree)
Change in Quality of Life Assessment | Baseline, week 6, week 12
  The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) - Scale: 1-5 (1 = very poor, 5 = very good)
Change in Symptom Severity - 1 | Baseline, week 6, week 12
  Generalized Anxiety Disorder 7 (GAD-7) - Scale: 0-3 (0 = not at all, 3 = nearly every day)
Change in Symptom Severity - 2 | Baseline, week 6, week 12
  Montgomery-Asberg Depression Rating Scale (MADRS) - Scale: 0-6 (0 = not at all, 6 = frequent/very much)
Change in Symptom Severity - 3 | Baseline, week 6, week 12
  Patient Health Questionnaire 9 (PHQ-9) - Scale: 0-3 (0 = not at all, 3 = nearly every day)

SECONDARY OUTCOMES:
Qualitative Information: Healthcare Providers | Week 12
  Healthcare providers who administered the e-psychotherapy for duration of project will be asked through focus groups questions surrounding the feasibility of providing the e-psychotherapy, how it compared to in-person psychotherapy with respect to time commitment, feelings of 'connectedness' to participant, and any perceived benefits/drawbacks to e-psychotherapy.
Qualitative Information: Personal, social, and cultural factors | Week 12
  In focus groups, participants will be asked questions regarding personal, social, and cultural factors (gender, sexuality, background, supportive resources, structural/social barriers, etc.) that could impact participant experience with e-psychotherapy. This will be extracted using an Interpretive Phenomenological Analysis (IPA) approach.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Ethics and Data Privacy: Only care providers involved in care of participant will have access to charts. Patients will only be identifiable by ID number on OPTT platform and real identity and consent forms will be stored locally in locked file cabinet and destroyed 5 years after study completion date. Only anonymized data will be provided to analysis team members.
  OPTT is HIPAA, PIPEDA and SOC-2 compliant and all servers and databases are hosted in AWS Canada cloud infrastructure which is managed by Medstack to assure all provincial and federal privacy and security regulations are met. OPTT will not collect any identifiable personal information or IP addresses for privacy purposes. OPTT will only collect anonymized metadata to improve its service quality and provide advanced analytics to the clinician team. All data is encrypted by OPTT and no employee has direct access to patient data. All encrypted backups are kept in the S3 storage that is dedicated to Queen's University.

REFERENCES:
- [Derived] Moghimi E, Stephenson C, Agarwal A, Nikjoo N, Malakouti N, Layzell G, O'Riordan A, Jagayat J, Shirazi A, Gutierrez G, Khan F, Patel C, Yang M, Omrani M, Alavi N. Efficacy of an Electronic Cognitive Behavioral Therapy Program Delivered via the Online Psychotherapy Tool for Depression and Anxiety Related to the COVID-19 Pandemic: Pre-Post Pilot Study. JMIR Ment Health. 2023 Dec 25;10:e51102. doi: 10.2196/51102. PMID 37993984
- [Derived] Alavi N, Yang M, Stephenson C, Nikjoo N, Malakouti N, Layzell G, Jagayat J, Shirazi A, Groll D, Omrani M, O'Riordan A, Khalid-Khan S, Freire R, Brietzke E, Gomes FA, Milev R, Soares CN. Using the Online Psychotherapy Tool to Address Mental Health Problems in the Context of the COVID-19 Pandemic: Protocol for an Electronically Delivered Cognitive Behavioral Therapy Program. JMIR Res Protoc. 2020 Dec 18;9(12):e24913. doi: 10.2196/24913. PMID 33290245
- See also: Publication — https://pubmed-ncbi-nlm-nih-gov.proxy.queensu.ca/33290245/